CLINICAL TRIAL: NCT01438190
Title: A Comparison Study of a Novel Stimulation Protocol With Metformin in Step-down Regimen and the Conventional Low Dose Step-up Protocol in Patients With Polycystic Ovary Syndrome Undergoing in Vitro Fertilization
Brief Title: Metformin in Step-down Regimen Versus Conventional Low Dose Step-up Protocol in Patients With PCOS Undergoing IVF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, MD, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09/2011
Record Dates: First submitted 2011-09-19; First posted 2011-09-22 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Infertility; PCOS
MeSH Terms: conditions — Infertility | interventions — Metformin; Gonadotropins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Metformin plus step-down protocol
  Interventions: Drug: Metformin, gonadotropins in step-down regimen
- Control (Active Comparator): Placebo and step-up protocol
  Interventions: Drug: Placebo, gonadotropins in step-up regimen

INTERVENTIONS:
Drug: Metformin, gonadotropins in step-down regimen — Metformin 850 mg cps, two cps daily for 12 weeks. gonadotropins 75IU f, step-down regimen, starting dose of 225 IU daily.
  Arms: Experimental
Drug: Placebo, gonadotropins in step-up regimen — Placebo cps, two cps daily. Gonadotropins 75IU f, step-up regimen, starting dose of 75 IU daily.
  Arms: Control

SUMMARY:
Because many women with Polycystic Ovary Syndrome (PCOS) are very sensitive to the use of gonadotropins, several strategies have been proposed to reduce the risk of Ovarian hyperstimulation syndrome (OHSS) and multiple pregnancies.

The low dose step-up protocol and the step-down protocols in PCOS patients have been described in literature.

The step-down regimen is designed to achieve the follicle stimulating hormone (FSH) threshold through a loading dose of FSH with a subsequent stepwise reduction as soon as follicular development is observed on ultrasound. On the contrary the step-up regimen is based upon the principle of a stepwise increase in FSH supply to determine the FSH threshold for follicular development. After commencement of gonadotropin administration, if follicle development is not observed on ultrasound after 1 week, an increase in the dose is recommended. Once follicle growth is observed, the same FSH dose is maintained until follicular selection is achieved.

Preliminary studies report that both step-up and step-down regimens achieve similar high rates of monofollicular development. However, the largest study published so far has shown that the step-up regimen is safer in terms of monofollicular development.

Recent data demonstrate that metformin administration in infertile PCOS patients who are at high-risk for OHSS reduces the incidence and severity of OHSS during gonadotropin ovarian stimulation in a step-down regimen for in vitro fertilization (IVF) programs.

The aim of the present study will be to compare the conventional low dose step-up protocol and the combined protocol consisting in metformin and gonadotropin step-down regimen.

ELIGIBILITY:
Inclusion Criteria:

* PCOS
* Infertility
* High responders

Exclusion Criteria:

* Poor responders
* Major medical conditions

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
OHSS rate | one month
  Ovarian hyperstimulation syndrome

SECONDARY OUTCOMES:
cancellation rate | one month
  rate of cancelled cycle for high risk of OHSS or low response
pregnancy rate | one month
live-birth rate | nine months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- "Pugliese" Hospital, Catanzaro, Italy